CLINICAL TRIAL: NCT06007638
Title: A Randomised Double-Blinded, Placebo-Controlled, Single and Multiple Ascending Dose, Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LY3876602 in Healthy Participants
Brief Title: A Single and Multiple Ascending Dose Study of LY3876602 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18734; J4K-MC-LALA (Other: Eli Lilly and Company); 2023-504838-21-00 (EU CTIS Number)
Record Dates: First submitted 2023-08-18; First posted 2023-08-23 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- LY3876602 (Experimental): Single ascending doses of LY3876602 administered intravenously (IV).
  Interventions: Drug: LY3876602
- Placebo (Placebo Comparator): Placebo administered IV.
  Interventions: Drug: Placebo
- LY3876602 Part B (MAD) (Experimental): Multiple ascending doses of LY3876602 will be administered intravenously (IV).
  Interventions: Drug: LY3876602
- Placebo: Part B (MAD) (Placebo Comparator): Placebo administered IV
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3876602 — Administered IV.
  Arms: LY3876602; LY3876602 Part B (MAD)
Drug: Placebo — Administered IV.
  Arms: Placebo; Placebo: Part B (MAD)

SUMMARY:
The aim of this study is to evaluate the safety, tolerability and PK of LY3876602 after administering it as single ascending doses and, following a data review, proceeding to multiple ascending doses in healthy participants. Blood tests will also be performed to check how much LY3876602 gets into the bloodstream and cerebrospinal fluid (CSF) and how long it takes the body to eliminate it.

Following the screening visit for Part A, the study will last up to approximately 20 weeks., and a subgroup of participants will consent to CSF collections The study will last up to approximately 28 weeks for Part B. All participants will consent to CSF collections.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are overtly healthy as determined by medical evaluation
* Have a body mass index with the range of 18 and less than or equal to (≤) 32 kilograms per square meter (kg/m²)
* Male or female participants of nonchildbearing potential

Exclusion Criteria:

* Have a family history, defined as a parent or first-degree relative, of genetic neurodegenerative disorders
* Have allergies to diphenhydramine, epinephrine, or methylprednisolone
* Have serious or unstable medical conditions,
* History of skin wounding within 14 days of screening or current skin infection
* Are unwilling to stop alcohol consumption 48 hours prior to each dosing
* Have active or latent tuberculosis
* Participants in the cohorts undergoing lumbar puncture have an allergy to local anesthetics

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to 28 weeks
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3876602 | Predose up to 28 weeks
  PK: AUC of LY3876602
PK: Maximum Observed Drug Concentration (Cmax) of LY3876602 | Predose up to 28 weeks
  PK: Cmax of LY3876602
PK: Half-life (t1/2) of LY3876602 | Predose up to 28 weeks
  PK: t1/2 of LY3876602

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- ICON Early Phase Services, LLC, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No